CLINICAL TRIAL: NCT00788775
Title: A Phase II Study of Nilotinib (AMN107) In TKI Resistant or Intolerant Patients With Metastatic Mucosal, Acral or Chronically Sun Damaged Melanoma
Brief Title: Nilotinib in TKI Resistant or Intolerant Patients With Metastatic Mucosal, Acral, or Chronically Sun Damaged Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Novartis (Industry)
Responsible Party: Principal Investigator, F. Stephen Hodi, MD, Melanoma Disease Center Director, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-244
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Mucosal Lentiginous Melanoma; Acral Melanoma; Melanoma
Keywords: nilotinib
MeSH Terms: conditions — Melanoma | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib (Experimental): Nilotinib was given at a dose of 400 mg orally daily (200 mg pills twice per day). Patients received treatment up to 12 months as long as they were receiving clinical benefit.
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib
  Other Names: Tasigna; AMN107

SUMMARY:
Given the poor prognosis and limited treatment options available for patients with mucosal or acral/lentiginous melanomas who develop metastatic disease, genetic discoveries of KIT mutations in these cancers present the need to test multi-targeted kinase inhibitors with potent KIT inhibitory activity in this patient population. Imatinib and other tyrosine kinase inhibitors (TKIs) have the potential to be effective in this patient population, but patients may develop resistance to treatment. Therefore, in this study, we propose to test nilotinib in patients with metastatic mucosal, acral, or chronically sun-damaged melanoma following treatment with another TKI.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the proportion of patients, with metastatic mucosal, acral, or chronically sun damaged melanomas, whose tumors have KIT aberrations, and who progressed or could not tolerate a KIT targeting tyrosine kinase inhibitor (TKI) (e.g. including but not limited to imatinib mesylate, sunitinib, or dasatanib), who are alive and without progression of disease four months after beginning treatment with nilotinib.

Secondary

* To determine early evidence of biologic and clinical activity by best overall response rate.
* To estimate time to progression of disease and overall survival.
* To determine the tolerability of nilotinib.
* To evaluate the use of FDG-PET scanning in determining early biologic response to therapy.
* To correlate c-kit mutational status and amplification status with response to therapy.
* To evaluate the feasibility of nilotinib.
* To evaluate the tolerability of nilotinib in patients with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically documented diagnosis of mucosal melanoma or acral melanoma or chronically sun damaged melanoma as evidenced by solar elastosis on pathology
* Patient's tumor with evidence for KIT mutation or amplification. Patient tumors that already have documented mutations or amplification do not have to have tissue submitted again for analysis to confirm eligibility
* Have failed, progressed, or not been able to tolerate other tyrosine kinase inhibitors including but not limited to imatinib mesylate, sunitinib or dasatinib treatment.
* At least one measurable site of disease
* ECOG Performance Status 0, 1 or 2
* Adequate organ function as outlined in the protocol
* Negative pregnancy test for female patients of childbearing potential

Exclusion Criteria:

* Patient has received any other investigational agents within 28 days of first day of study drug dosing unless the disease is rapidly progressing
* Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ
* Female patients who are pregnant or breast-feeding
* Patient has a severe and/or uncontrolled medical disease
* Patient has a rare hereditary problem of galactose intolerance, severe lactase deficiency or of glucose-galactose malabsorption
* Patient with electrolyte abnormality unless the level can be corrected to normal levels prior to initiating study drug
* Known brain metastasis
* Known chronic liver disease
* Patient has received chemotherapy within 4 weeks prior to study entry, unless the disease is rapidly progressing (6 weeks for nitrosourea or mitomycin-C)
* Patient previously received radiotherapy to 25% or greater of the bone marrow
* Patient had a major surgery within 2 weeks prior to study entry
* Impaired cardiac function
* QTc > 450msec on screening ECG
* Myocardial infarction within one year prior to starting nilotinib
* Other clinically significant heart disease
* Patients who are currently receiving treatment with any of the medications that have the potential to prolong QT interval
* Patients who are currently receiving Warfarin > 1mg/day
* Patient with any significant history of non-compliance to medical regimens or with the inability to grant reliable informed consent
* Prior therapy with nilotinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-01-23 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F. Stephen Hodi, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - The Angeles Clinic and Research Institute, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carvajal RD, Lawrence DP, Weber JS, Gajewski TF, Gonzalez R, Lutzky J, O'Day SJ, Hamid O, Wolchok JD, Chapman PB, Sullivan RJ, Teitcher JB, Ramaiya N, Giobbie-Hurder A, Antonescu CR, Heinrich MC, Bastian BC, Corless CL, Fletcher JA, Hodi FS. Phase II Study of Nilotinib in Melanoma Harboring KIT Alterations Following Progression to Prior KIT Inhibition. Clin Cancer Res. 2015 May 15;21(10):2289-96. doi: 10.1158/1078-0432.CCR-14-1630. Epub 2015 Feb 18. PMID 25695690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on January 23, 2009 and closed early in December 2011 due to slow accrual. Patients enrolled from 8 medical centers beginning March 2009 through June 2011.
Groups:
- No CNS Metastastic Cohort; CNS Metastatic Cohort: Nilotinib was given at a dose of 400 mg orally daily (200 mg pills twice per day). Patients received treatment up to 12 months as long as they were receiving clinical benefit. Patients were classified into two cohorts based upon presence or absence of measurable brain metastases.
Period: Overall Study
Arm/Group | No CNS Metastastic Cohort | CNS Metastatic Cohort
Started | 11 | 9
Treated | 11 | 8
Completed | 1 | 1
Not Completed | 10 | 8
Not completed — Progressive Disease | 8 | 6
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Patient Non-Compliance | 1 | 0
Not completed — Patient's measurable disease resected. | 1 | 0

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of treated patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | No CNS Metastastic Cohort | CNS Metastatic Cohort | Total
Number analyzed (Participants) | 11 | 8 | 19
Age, Continuous [Median (Full Range); unit: years] | 68 [55 to 82] | 60 [38 to 85] | 67 [38 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 8 | 19
Melanoma Type [Number; unit: participants]
  Acral | 3 | 3 | 6
  Mucosal | 6 | 4 | 10
  Chronically Sun-Damaged (CSD) | 2 | 1 | 3
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) PS: (PS0) Fully active, able to carry on all pre-disease performance without restriction (PS1) Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (PS2) Ambulatory and capable of all self-care but unable to carry out any work activities; Up and about >50% of waking hours
  Participants
    ECOG PS0 | 7 | 4 | 11
    ECOG PS1 | 4 | 4 | 8
    ECOG PS2 | 0 | 0 | 0
CNS Metastatic Status [Count of Participants; unit: Participants] — Central Nervous System (CNS)
  Participants
    CNS Metastaic: No | 11 | 0 | 11
    CNS Metastaic: Yes | 0 | 8 | 8

OUTCOME MEASURES:

1. Primary Outcome: 4-month Progression-Free Survival Rate
Description: 4-month progression-free survival rate was defined as the proportion of patients absent death or progression based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST) before 4 months. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment; Treatment continued for 12 months unless disease progression or unacceptable toxicity. Relevant for this endpoint was disease status at 4 months.
Population: The analysis dataset is comprised of treated patients.
Measure: Number (90% Confidence Interval); unit: proportion of patients
Arm/Group | No CNS Metastastic Cohort | CNS Metastatic Cohort
Number analyzed (Participants) | 11 | 8
proportion of patients | 0.27 [0.08 to 0.56] | 0.125 [0.006 to 0.47]

2. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 8 weeks on treatment and long-term every 3 months until first progression, death or lost to follow-up. Mean treatment duration was 5.5 months (range 0-45; no/with CNS mets 7.4m/ 3m).
Population: The analysis dataset is comprised of treated patients.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | No CNS Metastastic Cohort | CNS Metastatic Cohort
Number analyzed (Participants) | 11 | 8
months | 3.4 [0.9 to 5.5] | 2.4 [1.8 to 3.9]

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from study entry to death or date last known alive.
Time Frame: Patients were followed long-term every 3 months until first progression, death or lost to follow-up. Median survival follow-up was 16.2 months (90%CI 11.7-17.7 months; no/with CNS mets 16.2m/ 11.7m).
Population: The analysis dataset is comprised of treated patients.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | No CNS Metastastic Cohort | CNS Metastatic Cohort
Number analyzed (Participants) | 11 | 8
months | 14.2 [7.1 to NA] — The upper limit of the 90% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 4.3 [3.5 to 11.9]

4. Secondary Outcome: Best Overall Response
Description: Best overall response (BOR) on treatment was based on RECIST 1.0 criteria. For target lesions, complete response (CR) is complete disappearance of all target lesions and partial response (PR) is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. CR or PR confirmation required within 4 weeks. Progressive disease (PD) is at least a 20% increase in the sum LD of target lesions from smallest sum LD as reference or the appearance of one or more new lesions. Stable disease (SD) is neither meeting PR or PD. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions. CR is disappearance of all non-target lesions.
Time Frame: as for outcome 2
Measure: Number; unit: participants
Arm/Group | No CNS Metastastic Cohort | CNS Metastatic Cohort
Number analyzed (Participants) | 11 | 8
participants
  Complete Response | 0 | 0
  Partial Response | 2 | 0
  Stable Disease | 4 | 6
  Progressive Disease | 4 | 1
  Unevaluable | 1 | 1

ADVERSE EVENTS:
Time Frame: AE assessment was ongoing from the start of study drug and up to day 30 post-treatment. Mean treatment duration was 5.5 months (range 0-45; no/with CNS mets 7.4m/ 3m).
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. Other AEs were defined as events with treatment-attribution of possible, probable or definite and grades 1 or 2 per CTCAEv3.
Arm/Group | No CNS Metastastic Cohort | CNS Metastatic Cohort
Serious Adverse Events (participants affected / at risk) | 3/11 | 1/8
Other Adverse Events (participants affected / at risk) | 9/11 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No CNS Metastastic Cohort (N=11) | CNS Metastatic Cohort (N=8)
Hepatic-other (Hepatobiliary disorders) | 1 | 0
ALT, SGPT (Investigations) | 1 | 0
AST, SGOT (Investigations) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Lipase (Investigations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | No CNS Metastastic Cohort (N=11) | CNS Metastatic Cohort (N=8)
Abdomen, pain (Gastrointestinal disorders) | 1 | 0
Alkaline phosphatase (Investigations) | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0
ALT, SGPT (Investigations) | 1 | 0
Amylase (Investigations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
AST, SGOT (Investigations) | 1 | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bilirubin (Investigations) | 1 | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac-other (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Constitutional, other (General disorders) | 0 | 1
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Edema limb (General disorders) | 1 | 0
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Fatigue (General disorders) | 7 | 1
Fever w/o neutropenia (General disorders) | 1 | 0
Head/headache (Nervous system disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 1
Incontinence urinary (Renal and urinary disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Joint, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Lipase (Investigations) | 1 | 0
Metabolic/Laboratory-other (Investigations) | 1 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Neuropathy-sensory (Nervous system disorders) | 0 | 1
Ocular-other (Eye disorders) | 1 | 0
Pain-other (General disorders) | 1 | 0
Pleura, pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 | 0
Scalp, pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin, pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin-other (Skin and subcutaneous tissue disorders) | 2 | 0
Taste disturbance (Nervous system disorders) | 0 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No